CLINICAL TRIAL: NCT04679402
Title: Diaphragm Function and Diver Endurance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Pro00107090
Record Dates: First submitted 2020-12-17; First posted 2020-12-22 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Muscles
Keywords: Control of breathing; Diaphragm function; Gas channels; Blood gases
MeSH Terms: interventions — Air

STUDY DESIGN:
Intervention Model Description: Mixed model with repeated measures
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The only person who will know the breathing gas is the trial coordinator. Since carbon monoxide is a colorless, tasteless gas, the subject will be unaware of the group they are in. The gas labeling will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respiratory Muscle Training Breathing Low Dose Carbon Monoxide (Experimental): Carbon monoxide 200 ppm in air breathing during daily 30 minute inspiratory loading training sessions. Subjects will breathe the experimental gas through a mouthpiece with nose-clip in place.
  Interventions: Other: Carbon monoxide 200 ppm in air
- Respiratory Muscle Training Breathing Air (Sham Comparator): Air breathing during daily 30 minute inspiratory loading training sessions. Subjects will breathe air through a mouthpiece with nose-clip in place.
  Interventions: Other: Carbon monoxide 200 ppm in air

INTERVENTIONS:
Other: Carbon monoxide 200 ppm in air — Low dose carbon monoxide

SUMMARY:
This project will test the following hypotheses:

1. Training of the inspiratory muscles increases underwater endurance and reduces hypercapnia in divers.
2. Inspiratory muscle training while breathing low concentration carbon monoxide (200 ppm) for 30 minutes daily improves diaphragm performance to a greater degree than the same training breathing air.
3. Inspiratory muscle training increases hypercapnia ventilatory response (gain) in those individuals with a low gain.
4. Variability in oxygen (O2) and carbon dioxide (CO2) permeability of erythrocyte membranes is a determining factor in underwater exercise performance.

DETAILED DESCRIPTION:
The aims of this project are to: (1) test a method that could increase personal endurance and reduce excessive rise in blood carbon dioxide during underwater exercise in divers; and (2) understand the mechanisms by which red blood cells transport oxygen and carbon dioxide and their possible effects on exercise capacity. During underwater exercise, personal endurance capacity and elevated blood PCO2 are key parameters that affect a diver's safety and performance. Unlike exercise on dry land, hypercapnia often occurs during dives and can impair cognitive function and predispose the diver to central nervous system (CNS) oxygen toxicity and convulsions underwater. Some people intrinsically have low ventilatory chemosensitivity, and are more likely to develop hypercapnia during a dive. Lack of stamina may also be a mission-critical variable, and both endurance and the ability to control blood carbon dioxide depend on the respiratory muscle (mainly diaphragm) function, for which endurance capacity is related to mitochondrial number. Previous studies from our lab have demonstrated increased mitochondrial biogenesis with training while breathing a low, sub-toxic (200 ppm) level of carbon monoxide. In this study we will test the effect of daily respiratory muscle training with and without added carbon monoxide on respiratory muscle power, diaphragm thickness, respiratory muscle endurance and exercise endurance during a subsequent dive to 50 feet of sea water. Arterial PCO2 and lactic acid levels will be measured during exercise tests before and after training. Transport of O2 and CO2 through erythrocyte cell membranes occurs mostly through channels. Erythrocytes from volunteers in this study will be tested for O2 and CO2 permeability, and to correlate gas transport efficiency with exercise performance and blood PCO2.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers
* Non-smokers
* Range of hypercapnic ventilatory responses
* VO2peak ≥35 mL.kg-1.min-1 (males)
* ≥30 mL.kg-1.min-1 (females)

Exclusion Criteria:

* Pregnancy
* Cardiorespiratory disease, including hypertension
* Neuromuscular disease
* Anemia
* Hemoglobinopathy, including sickle cell disease and trait

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Underwater endurance change | Baseline, 6 weeks
  Endurance during continuous underwater exercise at a depth of 50 ft below the surface
Arterial PCO2 change | Baseline, 6 weeks
  Blood gases during and at end of exercise
Ventilatory chemosensitivity change | Baseline, 6 weeks
  Hypercapnic ventilatory response (VE.min-1.mmHg)

SECONDARY OUTCOMES:
Erythrocyte gas channel analysis | Baseline
  Stopped-flow analysis of O2 offloading from Hb of (a) intact RBCs, (b) Hb in hemolysate

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Moon, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT04679402/ICF_000.pdf